CLINICAL TRIAL: NCT04960579
Title: Open-Label, Multicenter, Phase 1 Study to Assess the Safety of P-BCMA-ALLO1 in Subjects With Relapsed / Refractory Multiple Myeloma (MM)
Brief Title: P-BCMA-ALLO1 Allogeneic CAR-T Cells in the Treatment of Subjects With Multiple Myeloma
Acronym: MM
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Poseida Therapeutics, Inc. (Industry)
Collaborators: Roche-Genentech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-BCMA-ALLO1-001; XO44788 (Other: Poseida Therapeutics, Inc. a Member of the Roche Group)
Record Dates: First submitted 2021-06-24; First posted 2021-07-14 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (18):
- P-BCMA-ALLO1 CAR-T cells (Arm S) (Experimental): Single weight-based IV administration of P-BCMA-ALLO1 following conditioning chemotherapy regimen S.
  Rimiducid may be administered as indicated.
  Interventions: Biological: P-BCMA-ALLO1 CAR-T cells; Drug: Rimiducid
- P-BCMA-ALLO1 CAR-T cells (Arm F) (Experimental): Single weight-based IV administration of P-BCMA-ALLO1 following conditioning chemotherapy regimen F.
  Rimiducid may be administered as indicated.
  Interventions: Biological: P-BCMA-ALLO1 CAR-T cells; Drug: Rimiducid
- P-BCMA-ALLO1 CAR-T cells (Arm N) (Experimental): Single weight-based IV administration of P-BCMA-ALLO1. Rimiducid may be administered as indicated.
  Interventions: Biological: P-BCMA-ALLO1 CAR-T cells; Drug: Rimiducid
- P-BCMA-ALLO1 CAR-T cells (Arm P1) (Experimental): Single weight-based IV administration of P-BCMA-ALLO1 following conditioning chemotherapy regimen P1.
  Rimiducid may be administered as indicated.
  Interventions: Biological: P-BCMA-ALLO1 CAR-T cells; Drug: Rimiducid
- P-BCMA-ALLO1 CAR-T cells (Arm P2) (Experimental): Single weight-based IV administration of P-BCMA-ALLO1 following conditioning chemotherapy regimen P2.
  Rimiducid may be administered as indicated.
  Interventions: Biological: P-BCMA-ALLO1 CAR-T cells; Drug: Rimiducid
- P-BCMA-ALLO1 CAR-T cells (Arm R) (Experimental): Single weight-based IV administration of P-BCMA-ALLO1 following conditioning chemotherapy regimen R.
  Rimiducid may be administered as indicated.
  Interventions: Biological: P-BCMA-ALLO1 CAR-T cells; Drug: Rimiducid
- P-BCMA-ALLO1 CAR-T cells (Arm RS) (Experimental): Single weight-based IV administration of P-BCMA-ALLO1 following conditioning chemotherapy regimen RS.
  Rimiducid may be administered as indicated.
  Interventions: Biological: P-BCMA-ALLO1 CAR-T cells; Drug: Rimiducid
- P-BCMA-ALLO1 CAR-T cells (Arm C) (Experimental): Cyclic weight-based IV administration of P-BCMA-ALLO1 following conditioning chemotherapy regimen C.
  Rimiducid may be administered as indicated.
  Interventions: Biological: P-BCMA-ALLO1 CAR-T cells; Drug: Rimiducid
- P-BCMA-ALLO1 CAR-T cells (Arm160) (Experimental): Single fixed dose IV administration of P-BCMA-ALLO1 following conditioning chemotherapy regimen S, P1, P1.5 or P2.
  Rimiducid may be administered as indicated.
  Interventions: Biological: P-BCMA-ALLO1 CAR-T cells; Drug: Rimiducid
- P-BCMA-ALLO1 CAR-T cells (Arm480) (Experimental): Single fixed dose IV administration of P-BCMA-ALLO1 following conditioning chemotherapy regimen S, P1, P1.5 or P2.
  Rimiducid may be administered as indicated.
  Interventions: Biological: P-BCMA-ALLO1 CAR-T cells; Drug: Rimiducid
- P-BCMA-ALLO1 CAR-T cells (Arm P1.5) (Experimental): Single weight-based IV administration of P-BCMA-ALLO1 following conditioning chemotherapy regimen P1.5.
  Rimiducid may be administered as indicated.
  Interventions: Biological: P-BCMA-ALLO1 CAR-T cells; Drug: Rimiducid
- P-BCMA-ALLO1 CAR-T cells (Arm RP1) (Experimental): Single weight-based IV administration of P-BCMA-ALLO1 following conditioning chemotherapy regimen RP1.
  Rimiducid may be administered as indicated.
  Interventions: Biological: P-BCMA-ALLO1 CAR-T cells; Drug: Rimiducid
- P-BCMA-ALLO1 CAR-T cells (Arm RP1.5) (Experimental): Single weight-based IV administration of P-BCMA-ALLO1 following conditioning chemotherapy regimen RP1.5.
  Rimiducid may be administered as indicated.
  Interventions: Biological: P-BCMA-ALLO1 CAR-T cells; Drug: Rimiducid
- P-BCMA-ALLO1 CAR-T cells (Arm RP2) (Experimental): Single weight-based IV administration of P-BCMA-ALLO1 following conditioning chemotherapy regimen RP2.
  Rimiducid may be administered as indicated.
  Interventions: Biological: P-BCMA-ALLO1 CAR-T cells; Drug: Rimiducid
- P-BCMA-ALLO1 CAR-T cells (Arm CP1) (Experimental): Cyclic weight-based IV administration of P-BCMA-ALLO1 following conditioning chemotherapy regimen CP1.
  Rimiducid may be administered as indicated.
  Interventions: Biological: P-BCMA-ALLO1 CAR-T cells; Drug: Rimiducid
- P-BCMA-ALLO1 CAR-T cells (Arm CP1.5) (Experimental): Cyclic weight-based IV administration of P-BCMA-ALLO1 following conditioning chemotherapy regimen CP1.5.
  Rimiducid may be administered as indicated.
  Interventions: Biological: P-BCMA-ALLO1 CAR-T cells; Drug: Rimiducid
- P-BCMA-ALLO1 CAR-T cells (Arm CP2) (Experimental): Cyclic weight-based IV administration of P-BCMA-ALLO1 following conditioning chemotherapy regimen CP2.
  Rimiducid may be administered as indicated.
  Interventions: Biological: P-BCMA-ALLO1 CAR-T cells; Drug: Rimiducid
- P-BCMA-ALLO1 CAR-T cells (Arm MP1.5) (Experimental): Single weight based IV administration of P-BCMA-ALLO1 and methotrexate following conditioning chemotherapy regimen MP1.5 Rimiducid may be administered as indicated
  Interventions: Biological: P-BCMA-ALLO1 CAR-T cells; Drug: Rimiducid; Drug: Methotrexate

INTERVENTIONS:
Biological: P-BCMA-ALLO1 CAR-T cells — Allogeneic BCMA-targeted chimeric antigen receptor (CAR) T-cell therapy
Drug: Rimiducid — Safety switch activator
Drug: Methotrexate — Anti-metabolite
  Arms: P-BCMA-ALLO1 CAR-T cells (Arm MP1.5)

SUMMARY:
Phase 1 study comprised of open-label, dose escalation, multiple cohorts of P-BCMA-ALLO1 allogeneic T stem cell memory (Tscm) CAR-T cells in subjects with relapsed / refractory Multiple Myeloma (RRMM).

DETAILED DESCRIPTION:
Phase 1/1b study: Phase 1 Part 1 is a weight-based dose escalation following a 3+3 design of dose-escalating cohorts. Phase 1 Part 2 includes administration at fixed doses. After enrollment, subjects may receive a lymphodepletion therapy regimen before administration of allogeneic CAR-T cells, administered as a single or multiple dose(s). Treated subjects will undergo serial measurements of safety, tolerability and response. Rimiducid may be administered as indicated. Phase 1b of the study will undergo further expansion of cohorts/arms from Phase 1 Parts 1 or 2 or an intermediate dose between cohort levels.

ELIGIBILITY:
Inclusion Criteria:

1. Must have signed written, informed consent.
2. Males or females, ≥18 years of age.
3. Must have a confirmed diagnosis of active MM.
4. Must have measurable MM.
5. Must have relapsed / refractory MM, having received treatment with a proteasome inhibitor, immunomodulatory agent (IMiD), and anti-CD38 therapy.
6. Must be willing to practice birth control from the time of Screening and throughout the first year of the study after P-BCMA-ALLO1 administration.
7. Must have a negative serum pregnancy test at Screening and a negative urine pregnancy test within 3 days prior to initiating the lymphodepletion therapy regimen (females of childbearing potential).
8. Must be at least 90 days since autologous stem cell transplant, if performed.
9. Must have adequate vital organ function within pre-determined parameters.
10. Must have recovered from toxicities due to prior therapies.
11. Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.

Exclusion Criteria:

1. Is pregnant or lactating.
2. Has inadequate venous access.
3. Has active hemolytic anemia, plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome, disseminated intravascular coagulation, leukostasis, or amyloidosis.
4. Has an active second malignancy (not disease-free for at least 5 years) in addition to MM, excluding low-risk neoplasms such as non-metastatic basal cell or squamous cell skin carcinoma.
5. Has active autoimmune disease.
6. Has a history of significant central nervous system (CNS) disease, such as stroke, epilepsy, etc.
7. Has an active systemic infection.
8. Has a history of hepatitis B, hepatitis C virus, human immunodeficiency virus (HIV), or human T-lymphotropic virus (HTLV) infection, or any immunodeficiency syndrome. Subjects with a history of treated hepatitis C can be enrolled if negative by Hepatitis C PCR on multiple occasions.
9. Is positive for cytomegalovirus (CMV) by PCR, CMV immunoglobulin M (IgM) antibody, or Coronavirus disease 2019 (COVID-19) by PCR.
10. Has New York Heart Association (NYHA) Class III or IV heart failure, unstable angina, or a history of myocardial infarction or significant arrhythmia.
11. Has any psychiatric or medical disorder that would preclude safe participation in and/or adherence to the protocol.
12. Has received prior allogeneic cellular therapy or gene therapy.
13. Has received anti-cancer medications within 2 weeks of the time of initiating conditioning LD therapy.
14. Has received monoclonal antibody therapy within 4 weeks of initiating conditioning LD therapy.
15. Has received immunosuppressive medications within 2 weeks of the time of administration of P-BCMA-ALLO1, and/or expected to require them while on study.
16. Has received systemic corticosteroid therapy within 1 week or 5 half-lives (whichever is shorter) of the administration of P-BCMA-ALLO1 or is expected to require it during the course of the study.
17. Has CNS metastases or symptomatic CNS involvement of their myeloma.
18. Has a history of severe immediate hypersensitivity reaction to any of the agents used in this study.
19. Has a history of having undergone allogeneic stem cell transplantation, or any other allogeneic or xenogeneic transplant, or has undergone autologous transplantation within 90 days.
20. Arms R, RS, RP1, RP1.5 and RP2 Only: a) Has received a live vaccine within the last 28 days of the first administration of agents used in Arm R or RS, b) Has any known hypersensitivity or severe reactions or toxicity to agents used in Arms R or RS.
21. Has received radiation within 1 week of initiating conditioning LD therapy.
22. Administration of a live vaccine within the last 28 days prior to administration of LD therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2042-03 (Estimated)

PRIMARY OUTCOMES:
Phase 1 Part 1: Assess the safety and maximum tolerated dose (MTD) of P-BCMA-ALLO1 based on dose limiting toxicities (DLT) | Baseline through Day 28
  Rate of dose limiting toxicities (DLT)
Phase 1 Part 2: Assess the safety and tolerability of P-BCMA-ALLO1 when administered as a fixed dose of cells. | Baseline through 36 months
  Frequency and severity of adverse events, including cytokine release syndrome.
Phase 1b: The effect of cell dose and study arm | Baseline through 36 months
  Overall response rate (ORR) based on International Myeloma Working Group (IMWG) uniform response criteria

SECONDARY OUTCOMES:
The safety of P-BCMA-ALLO1 | Baseline through 15 years
  Incidence and severity of treatment-emergent adverse events
The anti-myeloma effect of P-BCMA-ALLO1 (ORR) in Phase 1 Parts 1 and 2 | Baseline through 15 years
  According to the International Myeloma Working Group (IMWG) Uniform Response Criteria for Multiple Myeloma: Overall Response Rate (ORR) - Percentage of patients with complete response (CR), very good partial response (VGPR), or partial response (PR)
Safety and Efficacy (anti-myeloma effect) will be used to guide the selection of RP2D | Baseline through 15 years
  According to the International Myeloma Working Group (IMWG) Uniform Response Criteria for Multiple Myeloma: Time to Response (TTR) - Time to complete response (CR), very good partial response (VGPR), or partial response (PR) to progressive disease, Overall response rate (ORR), Duration of response (DOR), Progression free survival (PFS), and Overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Maika Onishi, M.D., Study Director — Senior Medical Director
Locations (22):
- United States (22):
  - City of Hope, Goodyear, Arizona
  - University of California San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia
  - Blood Marrow and Transplant Group of Georgia, Atlanta, Georgia
  - City of Hope, Chicago, Illinois
  - Advocate Aurora Health, Park Ridge, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Wayne State - Karmanos Cancer Institute, Detroit, Michigan
  - Hackensack Meridian Health, Hackensack, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma, Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Sarah Cannon Research Institute - St. David's South Austin Medical Center, Austin, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - Sarah Cannon Research Institute - Methodist Healthcare, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tseng H, Dholaria B, Cranert SA, Richter M, Marquez KS, Cho BS, Bacong A, McArthur K, Eskew JD, McCaigue J, Haag S, Krasny A, Solimine B, Coffey MJ, Loyola A, Kwong J, Shune L, Kin A, Costello CL, Kocoglu MH, Ramakrishnan A, Namini H, Martin CE, Belani R, Coronella J, Shedlock DJ. TSCM-predominant allogeneic anti-BCMA CAR-T therapy for relapsed/refractory multiple myeloma: preclinical characterization and interim results from a phase 1 trial. Nat Commun. 2025 Nov 24;16(1):10050. doi: 10.1038/s41467-025-65267-0. PMID 41285709